CLINICAL TRIAL: NCT03096964
Title: Effects of Nordic Walking Training in Energetic, Mechanical and Neuromuscular Parameters of Elderly. A Randomized Clinical Trail
Brief Title: Nordic Walking Training for Older People
Acronym: Pole walking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Leonardo A. Peyré-Tartaruga, Adjunct Professor, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LTartaruga,
Record Dates: First submitted 2016-12-08; First posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Sedentary Lifestyle; Age Problems
Keywords: Elderly training; Pole walking; Locomotor Rehabilitation Index; Self-selected speed of walking; Recovery
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nordic walking (Experimental): Experimental: Nordic walking Training The total period of training was composed by 8-week of walking with poles, three sessions per week. The cycles were divided into eight microcycles composed by three training sessions. Each training session took 60 min. Nordic walking aerobics training were used during the training period. These exercises were performed alternating volume and intensity. Exercise intensities were controlled using the cardiac monitor, and the zone was since 70% to 105% of the heart rate at the second ventilatory threshold. And volume was controlled using the time of the session.
  Interventions: Other: Nordic walking training
- Free Walking (Experimental): Experimental: Free walking Training The total period of training was composed by a 8-week cycles of walking without poles, with three sessions per week. The cycles were divided into eight microcycles composed by three training sessions. Each training session took 60 min. Free walking aerobics training were used during the training period. These exercises were performed alternating volume and intensity. Exercise intensities were controlled using the cardiac monitor, and the zone was since 70% to 105% of the heart rate at the second ventilatory threshold. And volume was controlled using the time of the session.
  Interventions: Other: Free walking training

INTERVENTIONS:
Other: Free walking training — The training period begin for both groups, will be comprised of eight weeks of duration, with frequency of three weekly sessions. Volume (session duration in minutes) and intensity (percentage of the heart rate at second threshold ) were the same for both groups, only differing in the use (NW) or not of the poles (FW). Each session will have of the Initial Part or warming-up, the Main Part and Final Part or cooling-down.
  Arms: Free Walking
Other: Nordic walking training — The training period begin for both groups, will be comprised of eight weeks of duration, with frequency of three weekly sessions. Volume (session duration in minutes) and intensity (percentage of the heart rate at second threshold ) were the same for both groups, only differing in the use (NW) or not of the poles (FW). Each session will have of the Initial Part or warming-up, the Main Part and Final Part or cooling-down.
  Arms: Nordic walking

SUMMARY:
Objective: to assess by means of a randomized clinical trial the effects of eight weeks of Nordic walking and free walking training on quality of life (QoL), static balance, dynamic variability, self-selected walking speed (SWS) and locomotor rehabilitation index (LRI), parameters of pendular mechanism [external (Wext), internal (Wint) and total mechanical work (Wtot), Recovery (R), Cost of Transport (C)], Electromyographic parameters (Average signal and co-contraction of the Anterior deltoid (AD), triceps brachii (TB), vastus lateralis (VL), biceps femoris (BF), anterior tibial (AT) and medial gastrocnemius (MG) muscles, heart rate of exercise (HRexercise) - and the rate of perceived exertion (RPE), in sedentary elderly.

DETAILED DESCRIPTION:
Introduction: Considering the increase in the elderly population and their life expectancy, together with the expansion of Nordic walking (NW) interventions as a training method for the elderly, there is a need of preventive studies of RCTs and with methodological good quality approach to enable physical education, health and rehabilitation professionals to make decisions regarding the type, the volume and the intensity of NW exercise in promoting the health of the sedentary elderly. Objectives: The aim of this study is to evaluate, through a randomized clinical trial, the effects of eight weeks of NW and FW training on quality of life (QoL), static balance, dynamic variability, self-selected treadmill walking speed (SSWSTreadmill), Locomotor rehabilitation (LRI) Parameters of Pendular Mechanism (external, internal and total mechanical work -Wext, Wint, Wtot, Recovery -R,Cost of Transport - C), Electromyographic parameters (Average signal and co-contraction of the AD, TB, VL, BF, AT and MG muscles), heart rate of exercise - HRexercise and the rate of perceived exertion (RPE), in sedentary elderly. of sedentary elderly. Experimental Design: Randomized Controlled Clinical Trial (RCT). Study Site: School of Physical Education, Physiotherapy and Dance (ESEFID), Federal University of Rio Grande do Sul Porto Alegre, Rio Grande do Sul, Brazil. Methods: The sample comprised 33 sedentary participants randomly divided into two groups (Nordic walking group and Free walking group who will perform training for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary elderly people
* Aged between 60 and 80

Exclusion Criteria:

* Smoking
* Show chronic pain or presence of migraine or nausea in daily life;
* History of labyrinthitis

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Self-selected walking speed - SSWS | Change from baseline SSWS at 8 weeks
  This outcome will be measure through sub-maximal test of walking treadmill, using the portable gas analyser Equipment.

SECONDARY OUTCOMES:
Quality of life (QoL) | Change from baseline QoL at 8 weeks
  The quality of life will be estimated using the World Health Organization Quality of Life Project for elderly people (WHOQOL) instrument.
Locomotor rehabilitation index (LRI) | Change from baseline LRI at 8 weeks
  This outcome will be measure through of the measure on sub-maximal test of walking treadmill, using the three-dimensional motion analysis system (VICON).
Oxygen consumption (VO2) | from baseline to 8 weeks
  This outcome will be measure through of the of the walking test on treadmill and too using the portable gas analyzer equipment (units in ml/kg/min).
Cost of transport (C) | from baseline to 8 weeks
  This outcome will be measured through of the walking test on a treadmill will be collected the oxigem consumption using the portable gas analyzer equipment (measure unit in ml.O2.km).
Optimal Walking Speed (OPT) | from baseline to 8 weeks
  This outcome will be measure through of the registered image movement analysis using the three-dimensional motion analysis system (VICON) of the walking test on treadmill (unit in km/h)
Oxygen Consumption at anaerobic threshold (VO2VT2) | from baseline to 8 weeks
  This outcome will be measure through maximal progressive treadmill test, using the portable gas analyser VO2000 equipment.
Peak Oxygen Consumption (VO2peak) | from baseline to 8 weeks
  This outcome will be measure through maximal progressive treadmill test, using the portable gas analyser VO2000 equipment.
Heart Rate at anaerobic threshold (HRVT2) | from baseline to 8 weeks
  This outcome will be measure through maximal progressive treadmill test, using a heart rate monitor (POLAR, FT1).
Rest Heart Rate (HRrest) | from baseline to 8 weeks
  This outcome will be measure using a heart rate monitor (POLAR, FT1). The participants will remain seated in a quiet and controlled temperature room during 15 minutes prior to measurement of the heart rate.
Exercise Heart Rate (HRexercise) | from baseline to 8 weeks
  This outcome will be measure using a heart rate monitor (POLAR, FT1) measurement of the heart rate of exercise during the walking test on treadmill at different speed.
Rest Arterial Systolic Blood Pressure (SBPrest) | from baseline to 8 weeks
  This outcome will be measured through blood pressure ambulatory monitor (Meditech). The participants will remain seated in a quiet and controlled temperature room during 15 minutes prior to measurement of the arterial systolic blood pressure.
Rest Arterial Diastolic Blood Pressure (DBPrest) | Change from baseline DBPrest at 8 weeks
  This outcome will be measured through blood pressure ambulatory monitor (Meditech, ABPM-04 equipment). The participants will remain seated in a quiet and controlled temperature room during 15 minutes prior to measurement of the arterial systolic blood pressure.
Parameters of Static balance (Amplitude ans Speed of Center of pressure in X, Y and Z axis) | Change from baseline Parameters of Static Balance at 8 weeks
  This outcome will be measure through of Static Balance in Force Platform (AMTI)
Parameters of Dynamic variability (coefficient of variation (CoV) of Stride length (SL), stride frequency (SF), swing time (ST), and contact time (CT) | Change from baseline Parameters of Dynamic Balance at 8 weeks
  This outcome will be measure through of the variability on sub-maximal test of walking treadmill, using the three-dimensional motion analysis system (VICON).
Spatial Temporal Parameters (stride frequency, stride length, swing time and contact time) | Change from baseline Spatial Temporal parameters at 8 weeks
  This outcome will be measure through of the registered image movement analysis using the three-dimensional motion analysis system (VICON) of the walking test on treadmill at different speed of walking (1,2,3,4 and 5 km/h), 5 minutes at each speed.
Parameters of Pendular Mechanism (external, internal and total mechanical work, Wext, Wint and Wtot, respectively, Recovery). | Change from baseline Parameters of Mechanical Work at 8 weeks
  This outcome will be measure through of the registered image movement analysis using the three-dimensional motion analysis system (VICON) of the walking test on treadmill at different speed of walking (1,2,3,4 and 5 km/h), 5 minutes at each speed.
Other Parameters of Pendular Mechanism (Percentage of congruity (%Cong), instantaneous pendular transduction and Recovery of step, shift phase (PhaseShift). | Change from baseline other Parameters of Pendular Mechanism at 8 weeks
  This outcome will be measure through of the registered image movement analysis using the three-dimensional motion analysis system (VICON) of the walking test on treadmill at different speed of walking (1,2,3,4 and 5 km/h), 5 minutes at each speed.
Movement Body Center of Mass (BCoM) on X, Y, Z axis | Change from baseline of BCoM at 8 weeks
  This outcome will be measure through of the registered image movement analysis using the three-dimensional motion analysis system (VICON) of the walking test on treadmill at different speed of walking (1,2,3,4 and 5 km/h), 5 minutes at each speed.
Maximal voluntary contractions (MVC) of the muscles: anterior deltoid (AD), triceps brachii (TB), vastus lateralis (VL), biceps femoris (BF), anterior tibial (AT) and medial gastrocnemius (MG) | Change from baseline MVC at 8 weeks
  This outcome will be measured through Measuring the electromyographic activation during treadmill walking tests using the Miotool electromyograph
Electromyographic Parameters (mean amplitude of the signal and co-contraction) of the muscles: anterior deltoid (AD), triceps brachii (TB), vastus lateralis (VL), biceps femoris (BF), anterior tibial (AT) and medial gastrocnemius (MG) | Change from baseline Electromyographic parameters at 8 weeks
  This outcome will be measured through Measuring the electromyographic activation during treadmill walking tests using an electromyograph

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo A Peyré-Tartaruga, PhD, Principal Investigator — PhD student of the Federal University of Rio Grande do Sul- Brasil
Locations (1):
- Federal University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomenuka NA, Oliveira HB, da Silva ES, Passos-Monteiro E, da Rosa RG, Carvalho AR, Costa RR, Rodriguez Paz MC, Pellegrini B, Peyre-Tartaruga LA. Nordic walking training in elderly, a randomized clinical trial. Part II: Biomechanical and metabolic adaptations. Sports Med Open. 2020 Jan 13;6(1):3. doi: 10.1186/s40798-019-0228-6. PMID 31932999
- [Derived] Gomenuka NA, Oliveira HB, Silva ES, Costa RR, Kanitz AC, Liedtke GV, Schuch FB, Peyre-Tartaruga LA. Effects of Nordic walking training on quality of life, balance and functional mobility in elderly: A randomized clinical trial. PLoS One. 2019 Jan 30;14(1):e0211472. doi: 10.1371/journal.pone.0211472. eCollection 2019. PMID 30699211